CLINICAL TRIAL: NCT03004846
Title: A Two-part Trial to Evaluate the Safety, Tolerability, Clinical Effect and Systemic Exposure Potential of Topically Applied GSK2981278 Ointment in Subjects With Plaque Psoriasis
Brief Title: A Study of GSK2981278 Ointment in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203820; 2016-002671-10 (EudraCT Number)
Record Dates: First submitted 2016-12-02; First posted 2016-12-29 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
Keywords: Vehicle- controlled; GSK2981278; Plaque psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: GSK2981278 4% (Experimental): Subjects will receive topical application of GSK2981278 4% ointment twice daily for 8 weeks. Based on new safety information, the concentration of GSK2981278 may be lowered to 2% or 0.8%.
  Interventions: Drug: GSK2981278 ointment
- Part B: GSK2981278 4% and vehicle (Experimental): In Part B, subjects will receive topical application of GSK2981278 4 % ointment or vehicle ointment twice daily for 8 weeks. Based on new safety information, the concentration of GSK2981278 may be lowered to 2% or 0.8%.
  Interventions: Drug: GSK2981278 ointment; Drug: Vehicle ointment

INTERVENTIONS:
Drug: GSK2981278 ointment — GSK2981278 ointment will be applied topically twice daily for 8 weeks to all subjects in Part A and to randomized subjects in Part B. GSK2981278 will be a white to off-white ointment and a thin layer will be applied to all affected areas for given timeframe.
  GSK2981278 is available as white to off-white ointment in unit strength 4% (w/w), 2% (w/w) and 0.8% (w/w), for topical application for application as thin layer to all affected areas .
Drug: Vehicle ointment — It will be supplied as white to off-white vehicle ointment for topical application.
  Arms: Part B: GSK2981278 4% and vehicle

SUMMARY:
GSK2981278 is an inverse agonist of retinoic acid receptor-related orphan receptor (ROR) gamma. The aim of this study is to evaluate the safety, tolerability, clinical effect, and systemic exposure potential of topically applied GSK2981278 ointment in subjects with plaque psoriasis by treating all plaques on the body for 8 weeks. This single-center study will be conducted in two parts. Part A will be an open-label, single arm study and part B will be a double-blind, randomized, 2-arm, parallel-group, vehicle-controlled study. In Part A, 8 adult subjects and in Part B, 18 adult subjects with chronic stable plaque psoriasis will be enrolled. Total duration of study will be approximately 14 weeks. The results of this study will provide preliminary information about safety and efficacy of the drug and will help in providing the guidance for further development strategy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above, at the time of signing the informed consent.
* Subjects with clinical diagnosis of stable plaque psoriasis for more than or equal to 6 months, as confirmed by the investigator.
* BSA involvement more than or equal to 5 percent and less than or equal to 15 percent, excluding face and intertriginous areas, at Screening and Baseline. The area of psoriasis involvement may include up to 2 percent of total BSA on the scalp with only sparse terminal hair and/or vellus hair.
* A PGA score of greater than or equal to 2 at Baseline.
* One target plaque located on the trunk or proximal parts of extremities (excluding scalp, knees, and elbows) that is at least 9 Centimeter ^2 in size at Screening and Baseline with a TPSS greater than or equal to 5 and induration sub score greater than or equal to 2.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 2 weeks after the last dose of study medication: a) Vasectomy with documentation of azoospermia. The documentation on male sterility can come from the site personnel's: review of subject's medical records, medical examination and/or semen analysis, or medical history interview. B) Male condom. The allowed method of contraception is only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Female of non-reproductive potential (FNRP) is eligible to participate in this study if she meets at least one of the following conditions: a) Females with one of the following procedures documented and no plans to utilize assisted reproductive techniques (e.g., in vitro fertilization or donor embryo transfer): bilateral tubal ligation or salpingectomy, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, bilateral Oophorectomy (surgical menopause); b) Post-menopausal women including Females 60 years of age or older, A practical definition accepts menopause after 1 year without menses with an appropriate clinical profile, e.g., age appropriate, more than 45 years, in the absence of hormone replacement therapy (HRT) or medical suppression of the menstrual cycle (e.g., leuprolide treatment). In questionable cases for women less than 60 years of age, a blood sample with simultaneous follicle stimulating hormone and estradiol falling into the central laboratory's post-menopausal reference range is confirmatory (these levels need to be adjusted for specific laboratories/assays. Females fewer than 60 years of age, who are on HRT and wish to continue, and whose menopausal status is in doubt, should not be enrolled in this study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can enroll into the study and resume use of HRT.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Psoriasis other than plaque variant (i.e. acute psoriasis guttate, psoriasis punctata, psoriasis erythroderma or pustular psoriasis).
* Current evidence of another ongoing or any acute cutaneous infection, history of repeated or chronic significant skin infections (unless irrelevant in the opinion of the investigator, i.e. onychomycosis, labial herpes or other minor diagnosis).
* Clinically-relevant skin disease or other skin pathologies, that may, in the opinion of the investigator, contraindicate participation or interfere with skin evaluations.
* ALT more than 2x Upper limit of normal (ULN) and bilirubin more than 1.5x ULN (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval using Bazett's formula (QTcB) more than 450 milliseconds (msec) or QTcB more than 480 msec in subjects with Bundle Branch Block. The QTcB should be based on single QTcB values of ECG obtained over a brief recording period. If QTcB is outside the threshold value, triplicate ECGs may be performed with the QTcB values averaged.
* Any condition that, in the judgment of the investigator, would put the subject at un-acceptable risk for the participation in the trial.
* History of malignancy within 5 years prior to dosing, except adequately treated non-invasive cancer of the skin (basal or squamous cell).
* Use of prohibited concomitant medications or products within the defined periods before the Day 1 visit and during the trial
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Symptoms of a clinically significant illness that may, in the opinion of the investigator, influence the outcome of the trial in the 4 weeks before baseline visit and during the trial.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* For Part B only-the subject has participated in Part A of this study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 4 weeks, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Prolonged exposure to natural or artificial sources of ultraviolet (UV) radiation (e.g., exposure to sunlight other than that associated with usual daily activities, use of tanning booth, etc.) within 2 weeks prior to the Day 1 visit or intention to have such exposure during the study, thought by the investigator likely to modify the subject's psoriasis.
* In the opinion of the investigator or physician performing the initial examination the subject should not participate in the clinical trial, e.g. due to probable noncompliance, inability to understand the trial and give adequately informed consent, or inability to complete the Psoriasis Symptom Diary.
* Close affiliation with the investigator (e.g. a close relative) or persons working at bioskin GmbH or subject is an employee of sponsor.
* Subject is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic stable plaque psoriasis were recruited in this 2 part study to evaluate safety, tolerability and clinical effect of GSK2981278.
Pre-assignment Details: A total of 10 participants were screened; of which two were screen failures and eight were included in the treatment phase of Part A and received GSK2981278 4% ointment for 8 weeks. Part B of this study was not conducted as pre-defined efficacy criteria for continuing to Part B were not met. Hence no participants were enrolled in Part B.
Groups:
- GSK2981278 4%: Part A: Participants received 4% ointment of GSK2981278 twice daily for 8 weeks.
- GSK2981278 4%: Part B: Randomized participants were planned to receive 4% ointment of GSK2981278 twice daily for 8 weeks.
- Vehicle Ointment: Part B: Randomized participants were planned to receive vehicle ointment twice daily for 8 weeks.
Period: Part A (Up to 14 Weeks)
Arm/Group | GSK2981278 4%: Part A | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B (Up to 14 Weeks)
Arm/Group | GSK2981278 4%: Part A | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part B of this study was not conducted as pre-defined efficacy criteria for continuing to Part B were not met. Hence no participants were enrolled in Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2981278 4%: Part A | GSK2981278 4%: Part B | Vehicle Ointment: Part B | Total
Number analyzed (Participants) | 8 | 0 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (9.43) |  |  | 54.9 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 8 |  |  | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European heritage | 8 |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-treatment Serious Adverse Events (SAEs) and Non-SAEs: Part A
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. The analysis was performed on Safety analysis Population which comprised of all participants exposed to at least 1 application of study medication.
Time Frame: Up to Day 57
Population: Safety analysis Population
Measure: Number; unit: Participants
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Participants
  non-SAEs | 1
  SAEs | 0

2. Primary Outcome: Number of Participants With Application Site Tolerability Assessment Score During Treatment Period: Part A
Description: The investigator assessed application site tolerability focusing on the treated non-lesional skin surrounding the plaques at each visit using the 5-point tolerability assessment scale ranging from 0 (no intolerance) to 4 (very severe intolerance). Number of participants in the corresponding score at Day 1, 15, 29 and 57 has been presented.
Time Frame: Day 1, Day 15, Day 29, Day 57
Population: Safety analysis Population
Measure: Number; unit: Participants
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Participants
  Day 1; Grade 0 | 8
  Day 1; Grade 1 | 0
  Day 1; Grade 2 | 0
  Day 1; Grade 3 | 0
  Day 1; Grade 4 | 0
  Day 15; Grade 0 | 8
  Day 15; Grade 1 | 0
  Day 15; Grade 2 | 0
  Day 15; Grade 3 | 0
  Day 15; Grade 4 | 0
  Day 29; Grade 0 | 8
  Day 29; Grade 1 | 0
  Day 29; Grade 2 | 0
  Day 29; Grade 3 | 0
  Day 29; Grade 4 | 0
  Day 57; Grade 0 | 8
  Day 57; Grade 1 | 0
  Day 57; Grade 2 | 0
  Day 57; Grade 3 | 0
  Day 57; Grade 4 | 0

3. Primary Outcome: Number of Participants With Negative Urinalysis Results: Part A
Description: Urine samples were collected from participants to evaluate urinalysis parameters including glucose, protein, erythrocytes and ketones. Number of participants with negative or normal urinalysis results at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values.
Time Frame: Up to Day 57
Population: Safety analysis Population
Measure: Number; unit: Participants
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Participants
  Glucose; Baseline | 8
  Glucose; Day 15 | 8
  Glucose; Day 29 | 8
  Glucose; Day 57 | 8
  Protein; Baseline | 8
  Protein; Day 15 | 8
  Protein; Day 29 | 8
  Protein; Day 57 | 8
  Erythrocytes; Baseline | 8
  Erythrocytes; Day 15 | 8
  Erythrocytes; Day 29 | 8
  Erythrocytes; Day 57 | 8
  Ketones; Baseline | 8
  Ketones; Day 15 | 8
  Ketones; Day 29 | 8
  Ketones; Day 57 | 8

4. Primary Outcome: Change From Baseline in Potential of Hydrogen (pH) of Urine: Part A
Description: The pH scale measures how acidic or basic a substance is. The pH scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic. A pH greater than 7 is basic. Urine samples were collected from participants and urine pH levels were assessed at Baseline, Day 15, Day 29 and Day 57. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Scores on a scale
  Day 15 | 0.1 (0.83)
  Day 29 | -0.1 (0.35)
  Day 57 | -0.1 (0.35)

5. Primary Outcome: Change From Baseline in Specific Gravity of Urine: Part A
Description: Urine samples were collected from participants and specific gravity levels were assessed at Baseline, Day 15, Day 29 and Day 57. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Ratio
  Day 15 | 0.0019 (0.00799)
  Day 29 | 0.0019 (0.00530)
  Day 57 | 0.0025 (0.00707)

6. Primary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN), Glucose, Potassium, Sodium and Calcium Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including BUN, glucose, potassium, sodium and calcium. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (Mmol/L)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Millimoles per liter (Mmol/L)
  BUN; Day 15 | -0.2678 (1.23300)
  BUN; Day 29 | -0.3570 (0.42670)
  BUN; Day 57 | 0.4909 (1.40146)
  Glucose; Day 15 | 0.041632 (0.7296677)
  Glucose; Day 29 | 0.104081 (0.7258495)
  Glucose; Day 57 | 0.298366 (0.4163911)
  Potassium; Day 15 | -0.14 (0.272)
  Potassium; Day 29 | 0.00 (0.312)
  Potassium; Day 57 | 0.13 (0.328)
  Sodium; Day 15 | -1.1 (2.17)
  Sodium; Day 29 | 0.8 (2.25)
  Sodium; Day 57 | -0.4 (1.06)
  Calcium; Day 15 | 0.021 (0.0624)
  Calcium; Day 29 | 0.038 (0.0765)
  Calcium; Day 57 | -0.013 (0.0886)

7. Primary Outcome: Change From Baseline in Creatinine, Total and Direct Bilirubin Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including creatinine, total and direct bilirubin. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Micromoles per liter (µmol/L)
  Creatinine; Day 15 | -5.8565 (2.16212)
  Creatinine; Day 29 | -3.8675 (6.32075)
  Creatinine; Day 57 | -3.7570 (6.92444)
  Total bilirubin; Day 15 | 1.425 (2.7396)
  Total bilirubin; Day 29 | 1.995 (2.5171)
  Total bilirubin; Day 57 | -0.342 (1.4307)
  Direct bilirubin; Day 15 | 0.3705 (0.66154)
  Direct bilirubin; Day 29 | 0.3990 (0.79963)
  Direct bilirubin; Day 57 | 0.0000 (0.52706)

8. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including AST, ALT and alkaline phosphatase. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
International unit per liter (IU/L)
  AST; Day 15 | 1.3 (4.43)
  AST; Day 29 | -0.3 (2.92)
  AST; Day 57 | -0.3 (6.23)
  ALT; Day 15 | 2.8 (8.75)
  ALT; Day 29 | 0.6 (5.26)
  ALT; Day 57 | 2.0 (8.59)
  Alkaline phosphatase; Day 15 | 2.1 (5.87)
  Alkaline phosphatase; Day 29 | 2.9 (12.89)
  Alkaline phosphatase; Day 57 | -0.8 (11.80)

9. Primary Outcome: Change From Baseline in Protein and Albumin Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including protein and albumin. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Grams per liter (g/L)
  Protein; Day 15 | 1.9 (2.90)
  Protein; Day 29 | -1.4 (2.83)
  Protein; Day 57 | 1.8 (3.65)
  Albumin; Day 15 | 1.4 (1.92)
  Albumin; Day 29 | 1.3 (1.67)
  Albumin; Day 57 | 1.0 (2.56)

10. Primary Outcome: Change From Baseline in Platelet, Leukocyte, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including platelets, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Groups:
- GSK2981278 4%:Part A: Participants received 4% ointment of GSK2981278 twice daily for 8 weeks.
Arm/Group | GSK2981278 4%:Part A
Number analyzed (Participants) | 8
10^9 cells/L
  Platelet; Day 15 | -3.6 (50.90)
  Platelet; Day 29 | -1.0 (28.98)
  Platelet; Day 57 | 0.1 (25.31)
  Leukocytes; Day 15 | 0.76 (2.745)
  Leukocytes; Day 29 | 0.42 (0.910)
  Leukocytes; Day 57 | 0.35 (0.780)
  Neutrophils; Day 15 | 0.695 (2.7477)
  Neutrophils; Day 29 | 0.144 (1.1659)
  Neutrophils; Day 57 | 0.217 (0.4432)
  Lymphocytes; Day 15 | -0.019 (0.6335)
  Lymphocytes; Day 29 | 0.243 (0.4457)
  Lymphocytes; Day 57 | 0.151 (0.3756)
  Monocytes; Day 15 | 0.090 (0.2778)
  Monocytes; Day 29 | -0.040 (0.2099)
  Monocytes; Day 57 | -0.063 (0.2344)
  Eosinophils; Day 15 | 0.019 (0.1579)
  Eosinophils; Day 29 | 0.085 (0.1321)
  Eosinophils; Day 57 | 0.029 (0.0825)
  Basophils; Day 15 | -0.008 (0.0287)
  Basophils; Day 29 | 0.001 (0.0264)
  Basophils; Day 57 | 0.004 (0.0151)

11. Primary Outcome: Change From Baseline in Erythrocyte Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including erythrocytes. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
10^12 cells/L
  Day 15 | 0.013 (0.2042)
  Day 29 | 0.055 (0.2555)
  Day 57 | 0.061 (0.2785)

12. Primary Outcome: Change From Baseline in Hemoglobin Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including hemoglobin. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
g/L
  Day 15 | 1.3 (6.18)
  Day 29 | 2.6 (7.63)
  Day 57 | 1.5 (9.18)

13. Primary Outcome: Change From Baseline in Hematocrit Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including hematocrit. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Proportion of Red blood cells in blood
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Proportion of Red blood cells in blood
  Day 15 | 0.0040 (0.01752)
  Day 29 | 0.0090 (0.02203)
  Day 57 | 0.0076 (0.02628)

14. Primary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV) Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCV. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Femtoliter (fL)
  Day 15 | 0.46 (1.235)
  Day 29 | 0.86 (1.112)
  Day 57 | 0.34 (1.172)

15. Primary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH) Levels: Part A
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCH. Change from Baseline in clinical hematology parameters at Day 15, Day 29 and Day 57 are presented. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Picograms (Pg)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Picograms (Pg)
  Day 15 | 0.16 (0.325)
  Day 29 | 0.21 (0.253)
  Day 57 | -0.06 (0.421)

16. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Levels: Part A
Description: Vital sign measurements including SBP and DBP were taken in a seated or supine position after 5-minutes of rest. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Millimeters of mercury (mmHg)
  SBP; Day 15 | -1.9 (4.58)
  SBP; Day 29 | -2.5 (4.63)
  SBP; Day 57 | -2.5 (2.67)
  DBP; Day 15 | 0.0 (2.67)
  DBP; Day 29 | 1.3 (4.43)
  DBP: Day 57 | 0.6 (4.17)

17. Primary Outcome: Change From Baseline in Pulse Rate Levels: Part A
Description: Vital sign measurements including pulse rate were taken in a seated or supine position after 5-minutes of rest. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Beats per minute
  Day 15 | 3.3 (9.19)
  Day 29 | 0.3 (12.21)
  Day 57 | 1.3 (11.36)

18. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters Including Single RR Heart Rate: Part A
Description: Single measurements of 12-lead ECG were obtained using an ECG machine to measure RR heart rate. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Beats per minute
  Day 29 | -2.5 (16.81)
  Day 57 | -3.5 (12.42)

19. Primary Outcome: Change From Baseline in ECG Parameters Including PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Bazett's Formula (QTcB) and RR Interval: Part A
Description: Single measurements of 12-lead ECG were obtained using an ECG machine to measure PR interval, QRS duration, QT interval, QTcB and RR interval. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value
Time Frame: Baseline and up to Day 57
Population: Safety analysis Population
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Milliseconds (msec)
  PR interval; Day 29 | -0.5 (9.78)
  PR interval; Day 57 | 7.3 (12.78)
  QRS duration; Day 29 | -0.5 (4.24)
  QRS duration; Day 57 | -0.3 (2.92)
  QT interval; Day 29 | 12.8 (28.88)
  QT interval; Day 57 | 9.0 (28.57)
  QTcB interval; Day 29 | 10.0 (15.62)
  QTcB interval; Day 57 | 3.5 (15.96)
  RR interval; Day 29 | 9.5 (170.62)
  RR interval; Day 57 | 13.0 (124.12)

20. Primary Outcome: Plasma Concentration of GSK2981278 at Nominal Time: Part A
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK2981278. Non-quantifiable values in a profile occurring before the first measurable concentration were assigned a value of zero concentration. Single non-quantifiable values occurring between measurable concentrations in a profile were omitted. The analysis was performed on PK analysis Population which comprised of participants with at least one sample collected and analyzed for plasma drug concentration. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10 hours post-dose on Day 1, Day 29 and Day 57; Pre-dose, 2 hours post-dose on Day 15
Population: PK analysis Population
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (Pg/mL)
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Picograms per milliliter (Pg/mL)
  Pre-dose; Day 1; n= 8 | 0.00 (0.000)
  1 hour post-dose; Day 1; n= 8 | 151.89 (210.535)
  2 hours post-dose; Day 1; n= 8 | 281.54 (589.927)
  4 hours post-dose; Day 1; n= 8 | 171.38 (160.357)
  6 hours post-dose; Day 1; n= 8 | 610.73 (1141.415)
  8 hours post-dose; Day 1; n= 8 | 192.06 (168.443)
  10 hours post-dose; Day 1; n= 8 | 554.94 (828.825)
  Pre-dose; Day 15; n= 7: number analyzed (Participants) | 7
  Pre-dose; Day 15; n= 7 | 1203.71 (1203.796)
  2 hours post-dose; Day 15; n= 8 | 893.00 (737.610)
  Pre-dose; Day 29; n= 8 | 1122.00 (587.760)
  1 hour post-dose; Day 29; n= 8 | 1299.63 (910.793)
  2 hours post-dose; Day 29; n= 8 | 1062.38 (662.050)
  4 hours post-dose; Day 29; n= 8 | 769.38 (369.861)
  6 hours post-dose; Day 29; n= 8 | 1022.63 (720.269)
  8 hours post-dose; Day 29; n= 7: number analyzed (Participants) | 7
  8 hours post-dose; Day 29; n= 7 | 897.71 (325.169)
  10 hours post-dose; Day 29; n= 8 | 875.38 (584.879)
  Pre-dose; Day 57; n= 8 | 875.75 (707.446)
  1 hour post-dose; Day 57; n= 8 | 1273.75 (784.902)
  2 hours post-dose; Day 57; n= 8 | 1077.00 (1128.070)
  4 hours post-dose; Day 57; n= 8 | 758.13 (494.661)
  6 hours post-dose; Day 57; n= 8 | 760.38 (550.695)
  8 hours post-dose; Day 57; n= 8 | 809.13 (373.947)
  10 hours post-dose; Day 57; n= 8 | 841.25 (579.772)

21. Primary Outcome: Number of Participants With SAEs and Non-SAEs: Part B
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. The analysis was performed on Safety analysis set Population which comprised of all participants exposed to at least 1 application of study medication. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to Day 57
Population: Safety analysis population. . Data was not collected for Part B as no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Number of Participants With Application Site Tolerability Assessment Score During Treatment Period: Part B
Description: The investigator planned to assess application site tolerability focusing on the treated non-lesional skin surrounding the plaques at each visit using the 5-point tolerability assessment scale ranging from 0 (no intolerance) to 4 (very severe intolerance). Number of participants with Application site tolerability assessment score were planned to be analyzed. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to Day 57
Population: Safety analysis Population. Data was not collected for Part B as no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Number of Participants With Change in Clinical Chemistry Toxicity Grade From Baseline: Part B
Description: Blood samples were planned to be collected for evaluation of clinical chemistry parameters. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as by subtracting post-Baseline visit values minus Baseline value. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Baseline and up to Week 57
Population: as for outcome 22
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Number of Participants With Change in Hematology Toxicity Grade From Baseline: Part B
Description: Blood samples were planned to be collected for the analysis of hematology parameters. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Baseline and up to Day 57
Population: as for outcome 22
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Number of Participants With Critical Changes in Values of Vital Signs in Response to Drug: Part B
Description: Vital sign measurement includes SBP, DBP, temperature, pulse rate. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to Day 57
Population: as for outcome 22
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Number of Participants With Abnormal Findings for ECG Parameters: Part B
Description: Single measurements of 12-lead ECGs were planned to be obtained using an ECG machine. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to Day 57
Population: as for outcome 22
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Mean Percent Change in TPSS From Baseline to Week 8: Part B
Description: The TPSS is the measure of clinical effect of GSK2981278. TPSS Total score was calculated by adding the individual scores of erythema, scaling, and induration (plaque thickness), assessed by the investigator on a 5-point scale ranging from 0=none to 4=very marked. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population. Data was not collected for Part B as no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Mean Percent Change in PGA Score From Baseline to Week 8: Part B
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. The 5-point scale ranges from 0=clear to 4=severe. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as by subtracting post-Baseline visit values minus Baseline value. Percent change from Baseline was calculated by dividing change from baseline value by Baseline value and multiplying it by 100. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population. Data was not collected for Part B as no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Mean Percent Change in PASI From Baseline to Week 8: Part B
Description: The PASI is a standard tool for assessing the severity of psoriasis that considers the overall severity of erythema, thickness, and scale, and the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=none to 4=severe) and the percent BSA affected is scored on a 7-point scale (0= 0% skin with psoriasis to 6=>=90% skin with psoriasis). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. Last observation values collected were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Percent change from Baseline was calculated by dividing change from baseline value by Baseline value and multiplying it by 100. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population. Data was not collected for Part B as no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part B | Vehicle Ointment: Part B
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Mean Percent Change From Baseline in Target Plaque Severity Score (TPSS): Part A
Description: The TPSS is the measure of clinical effect of GSK2981278. A target lesion of at least 9 centimeter square (cm^2) with a TPSS >=5 and an induration sub score >=2 was selected at Baseline. TPSS Total score was calculated by adding the individual scores of erythema, scaling, and induration (plaque thickness), assessed by the investigator on a 5-point scale ranging from 0=none to 4=very marked. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Percent change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplying it by 100. The analysis was performed on per protocol (PP) analysis Population which comprised of all participants eligible for treatment phase and who comply closely with the protocol.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Percent change
  Day 15 | -6.5 (7.24)
  Day 29 | -3.0 (5.74)
  Day 57 | -4.3 (10.61)

31. Secondary Outcome: Mean Percent Change From Baseline in Physician's Global Assessment (PGA) Score: Part A
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. The 5-point scale ranges from 0=clear to 4=severe. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Percent change from Baseline was calculated by dividing change from baseline value by Baseline value and multiplying it by 100.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Percent change
  Day 15 | -3.1 (8.84)
  Day 29 | -3.1 (8.84)
  Day 57 | 0.0 (0.0)

32. Secondary Outcome: Mean Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score: Part A
Description: The PASI is a standard tool for assessing the severity of psoriasis that considers the overall severity of erythema, thickness, and scale, as well as the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=none to 4=severe) and the percent BSA affected is scored on a 7-point scale (0= 0% skin with psoriasis to 6=>=90% skin with psoriasis) for each of the 4 specified body regions. The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. Last observation values collected prior to the first application of study treatment were considered as Baseline values. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Percent change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplying it by 100.
Time Frame: Baseline and up to Week 8
Population: PP analysis Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2981278 4%: Part A
Number analyzed (Participants) | 8
Percent change
  Day 15 | -3.98 (10.459)
  Day 29 | -0.27 (4.058)
  Day 57 | 4.26 (7.119)

ADVERSE EVENTS:
Time Frame: On-therapy SAEs and non-SAEs are presented from the start of study treatment up to Day 57.
Description: On-therapy SAEs and non-serious AEs are reported for members of the Safety analysis Population. Data was not collected for Part B because no Participants were enrolled into this part of the study.
Arm/Group | GSK2981278 4%: Part A | GSK2981278 4%: Part B | Vehicle Ointment: Part B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/8 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2981278 4%: Part A (N=8) | GSK2981278 4%: Part B (N=0) | Vehicle Ointment: Part B (N=0)
COMMON COLD (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03004846/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03004846/SAP_001.pdf